CLINICAL TRIAL: NCT01844193
Title: A 12-Month Prospective, Post-Market Study of Early Postoperative Compex® Rehab NMES Use in Total Knee Arthroplasty Patients
Brief Title: Early Postoperative Compex Rehab NMES Use for Total Knee Arthroplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Research Foundation (Other)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DJO-NMES-12
Record Dates: First submitted 2013-01-11; First posted 2013-05-01 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Therapy (No Intervention): This arm of the study will follow the standard therapy course after total knee arthroplasty.
- Standard Therapy + NMES (Experimental): This arm will follow the standard course of therapy but also incorporate daily neuromuscular electrical stimulation into the daily therapy regimen after total knee arthroplasty through use of the Compex Rehab device.
  Interventions: Device: Compex Rehab

INTERVENTIONS:
Device: Compex Rehab — Participants in this arm will use a Compex® Rehab unit for neuromuscular electrical stimulation starting with postoperative at-home day 1 and continue using the unit twice a day, every day, until a 10-week follow-up is reached. The unit produces a 380 microsecond biphasic curve and utilizes a four phase process for the treatment ("Warm-up", "Work", "Relaxation", and "Recovery") for a total treatment time of 20 minutes and 5 seconds per session. All frequencies are delivered at the maximum subjective tolerable intensity. Participants will control this intensity and be asked to select a level that is tolerable although mildly uncomfortable; they will be instructed to increase this intensity as tolerated.
  Arms: Standard Therapy + NMES

SUMMARY:
This study will examine the effects, if any, of using muscle stimulation on the quadriceps following a total knee replacement. Secondary objectives will be to evaluate and compare pain levels, qualitative outcomes, and the impact of NMES on pain medication requests between groups. It is possible that strengthening the quadriceps muscles and improving their activation will reduce postoperative pain and help patients return to activities sooner than with standard therapy alone.

DETAILED DESCRIPTION:
Neuromuscular electrical stimulation (NMES) for muscle strengthening and training has been in use since the 1970s, but questions still remain regarding its effectiveness with different patient populations, the duration of use and specifics regarding the stimulation itself, such as length and type of electrical impulse. NMES works by passing electrical impulses through the muscles to get them to contract. These impulses mimic the body's natural neural activity (action potential) to cause a contraction. The goal with NMES is to strengthen the muscle sooner by using muscle re-education. The quadriceps is weakened and sometimes slow to respond after knee surgery. A weak quadriceps muscle after surgery can be a contributing factor to dissatisfaction with the surgical result. When the quadriceps are weak or not firing properly, forces are transferred to areas such as the knee joint placing an additional strain on the replaced joint and contributing to knee pain, swelling and inflammation. If we can get patients' quads firing better and sooner, we hope we would also see better short-term and long-term functional outcomes and more long-term satisfaction than is presently reported. Study Enrollment We are looking for 60 patients to participate. We are randomly assigning 30 participants to receive the standard therapy regimen and 30 to follow the standard therapy regimen with the addition of using an NMES treatment twice a day, every day, for a ten-week period. Patients in the therapy with NMES treatment group will keep a tracking log of their use at home and will turn in the units at the 10-week appointment. The unit is easy to use and all participants are given specific instructions on its use. All participants complete baseline muscle testing before their surgery and then again at two-week, six-week, ten-week, and one-year appointments. The muscle testing consists of a battery of functional measures to assess the quadriceps such as the Timed Up and Go test (TUG), Six Minute Walk test (6MWT), Single Limb Stance (SLS) and others. All testing is conducted at Indiana Orthopaedic Hospital South's physical therapy department.

When designing this study we worked closely with the department to make sure the intended tests were appropriate both for our study and the facility; the input from the staff was and continues to be integral to this study's success. It is too early to report any findings and we are still enrolling patients. If effective, the NMES treatment should improve quadriceps activation and functioning early on after surgery, which will hopefully allow the patient to experience less pain and have a quicker functional recovery than a patient who did not use the NMES. Only time will tell if this is a logical conclusion and if NMES as a standard postoperative therapy would be beneficial for our patients. We anxiously await the outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for unilateral primary total knee arthroplasty and has a primary diagnosis of osteoarthritis.
* Patient is a male or non-pregnant female age 18 and older at time of surgery.
* Patient has signed an Institutional review board (IRB)-approved, study-specific informed consent form.
* Patient is willing and able to comply with the postoperative scheduled clinical evaluations and rehabilitation.

Exclusion Criteria:

* Patient has active infection within the affected knee joint.
* Patient requires revision surgery of a previously implanted total knee arthroplasty.
* Patient is morbidly obese, defined as having a body mass index (BMI) greater than or equal to 36.
* Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the intervention.
* Patient has been diagnosed with a systemic disease or current life threatening illness and is not able to carry on normal activities of daily life (e.g. Paget's disease, renal osteodystrophy, etc.).
* Patient has a history of cardiac issues including myocardial infarction and/or has a pacemaker.
* Patient is immunologically suppressed or receiving chronic steroids in excess of 5mg per day.
* Patient has a recent history of substance dependency that may result in deviations from the evaluation schedule.
* Patient is a prisoner.
* Patient has indication for contralateral total knee arthroplasty within the evaluation window.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Kolisek, MD, Principal Investigator — OrthoIndy South
Locations (1):
- OrthoIndy, Greenwood, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 patients were consented, but due to the gap between the consenting appointment and the baseline appointment, many patients failed to complete their baseline appointment or rescheduled/canceled their surgeries. Only patients attending the baseline appointment were considered enrolled.
Period: Overall Study
Arm/Group | Standard Therapy | Standard Therapy + NMES
Started | 19 | 21
Completed | 13 | 15
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy | Standard Therapy + NMES | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Full Range); unit: years] | 61 [51 to 72] | 62 [46 to 73] | 62 [46 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 9 | 14 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Quad Force [Mean (Full Range); unit: Newtons (N)] | 276.8 [147 to 479] | 291.1 [94 to 511] | 282.38 [94 to 511]

OUTCOME MEASURES:

1. Primary Outcome: Change in Quadriceps Force
Description: Change in quadriceps force is the difference between average quadriceps force measurements (in Newtons) obtained at the 1-year postoperative follow-up minus the average quadriceps force measurement at baseline. Averages are stratified by study arm. Negative values indicate a reduction in quadriceps force from baseline measurement to 1-year.
Time Frame: Baseline and 1-year Follow-up
Measure: Mean (Full Range); unit: Newtons (N)
Arm/Group | Standard Therapy | Standard Therapy + NMES
Number analyzed (Participants) | 19 | 21
Newtons (N) | 49.0 [-175.92 to 128.92] | 28.4 [-172.3 to 116.4]

2. Secondary Outcome: Change in VAS Pain Scores
Description: Average Visual Analog Scale (VAS) pain scores were computed for baseline and 1-year visits for each study arm. This measure is the difference between the average pain score at the baseline and 1-year follow-ups (1-year minus Baseline), stratified by study arm. The scale ranges from 0 to 10, with 0 being "No Pain" and 10 being " Pain as bad as it could possibly be." Lower scores indicate lower levels of reported pain. Negative scores indicate a reduction in pain from baseline to 1-year.
Time Frame: Baseline and 1-year Follow-up
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Standard Therapy | Standard Therapy + NMES
Number analyzed (Participants) | 19 | 21
score on a scale | -1.06 [-1.89 to -0.56] | -1.07 [-1.64 to -.056]

ADVERSE EVENTS:
Time Frame: Each subject was questioned about experiences of adverse events at each appointment after baseline and up until that subject completed their 1-year follow-up appointment. Should adverse event information have been reported after a subject completed their final study visit, but before study closeout, those data would also be included herein.
Arm/Group | Standard Therapy | Standard Therapy + NMES
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/21
Other Adverse Events (participants affected / at risk) | 2/19 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Therapy (N=19) | Standard Therapy + NMES (N=21)
Peptic Ulcer (Gastrointestinal disorders) | 0 | 1 — Patient reported checking into local Emergency Department due to concerns from seeing blood in stool.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=19) | Standard Therapy + NMES (N=21)
Knee Manipulation (Surgical and medical procedures) | 1 (1) | 0 (0)
Acid Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No